CLINICAL TRIAL: NCT02679118
Title: Evaluation of the Ability to Detect Bowel Gas During Laparoscopic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dan E. Azagury (Other)
Responsible Party: Sponsor-Investigator, Dan E. Azagury, Assistant Professor of Surgery, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: IRB-35295
Record Dates: First submitted 2016-02-04; First posted 2016-02-10 (Estimated); Last update posted 2017-08-18 (Actual); Status verified 2017-08

CONDITIONS: Intestinal Perforation
Keywords: intestinal perforation; bariatric surgery; gastric bypass; gastric perforation; colonic perforation
MeSH Terms: conditions — Intestinal Perforation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sentire (Experimental): The patients will undergo their laparoscopic gastric bypass, during the operative period at pre-defined time points, a small amount of gas from the abdomen will be withdrawn and analyzed for the device. The laparoscopic gastric bypass will proceed without interference or effect from the device.
  Interventions: Device: Sentire

INTERVENTIONS:
Device: Sentire — The device, at predetermined time points, will draw a small amount of gas from the abdomen. Upon obtaining the samples, the machine will analyze the sample for evidence of bowel gas. After each sample, the device will be purged prior to the acquisition of the next gas sample. The results of the analysis of the gas samples will be recorded for future analysis.

SUMMARY:
This study will determine the ability of the device to draw a small amount of gas from an insufflated abdomen during laparoscopic surgery and accurately detect if gaseous content from the bowel is present.

DETAILED DESCRIPTION:
Undetected bowel perforation is a rare but dangerous complication of laparoscopic surgery. If the injury is not detected and treated at the time of the surgical procedure, the patient can suffer sever complications including septic shock and eventually death. Our goal is to test a novel device that can detect bowel gas leakage from a perforation and alert the surgeon during the operation by evaluating the gases present in the insufflated abdomen during surgery. During laparoscopic surgery, carbon dioxide in inserted in the abdominal cavity in order to perform the operation. This is dynamic process as insufflation is a constant during the entire procedure to maintain a constant pressure and compensate small leaks due to the insertion and retrieval of instruments.

This study will determine the ability of device to be attached to a standard Veress needle or trocar during the operation and periodically draw a small amount of gas from the abdomen to evaluate the gas and accurately detect gaseous content from the bowel. Before the device can be used to detect bowel perforations, first we must ensure that it can accurately detect bowel gas in an insufflated abdomen.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 - 60 years old with the diagnosis of morbid obesity, who qualifies for laparoscopic gastric bypass surgical therapy, and has elected to undergo laparoscopic gastric bypass surgery.
2. Receiving care in the Stanford Hospital General Surgery Bariatric Surgery Clinic under the care of Dr. Dan Azagury
3. The patient is scheduled for laparoscopic roux en y gastric bypass surgery, with Dr. Azagury.
4. Willing and cognitively able to sign informed consent.

Exclusion Criteria:

1. Lack of or inability to provide informed consent.
2. Less than 18 years of age or greater than 60 years of age
3. Planned deviation from the standard laparoscopic gastric bypass operation
4. Conversion intra-operatively from a laparoscopic gastric bypass to an alternative laparoscopic surgical operation or to an open gastric bypass operation.
5. Enrollment in another device or drug study that may confound results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-02; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Methane levels released in the abdominal cavity from small bowel | Intra-operative measurement only
  Ability to detect and measure the level of methane released in the abdominal cavity by open small bowel
Hydrogen levels released in the abdominal cavity from small bowel | Intra-operative measurement only
  Ability to detect and measure the level of hydrogen released in the abdominal cavity by open small bowel

CONTACTS AND LOCATIONS:
Overall Officials: Dan Azagury, MD, Principal Investigator — Assistant Professor of Surgery
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Deffieux X, Ballester M, Collinet P, Fauconnier A, Pierre F; French National College of Gynaecologists and Obstetricians. Risks associated with laparoscopic entry: guidelines for clinical practice from the French College of Gynaecologists and Obstetricians. Eur J Obstet Gynecol Reprod Biol. 2011 Oct;158(2):159-66. doi: 10.1016/j.ejogrb.2011.04.047. Epub 2011 May 31. PMID 21621318
- [Background] Sahakian AB, Jee SR, Pimentel M. Methane and the gastrointestinal tract. Dig Dis Sci. 2010 Aug;55(8):2135-43. doi: 10.1007/s10620-009-1012-0. Epub 2009 Oct 15. PMID 19830557
- [Background] van der Voort M, Heijnsdijk EA, Gouma DJ. Bowel injury as a complication of laparoscopy. Br J Surg. 2004 Oct;91(10):1253-8. doi: 10.1002/bjs.4716. PMID 15376204